CLINICAL TRIAL: NCT05999708
Title: A Randomized, Double-Blind, Placebo-Controlled, Single, Repeat Dose Escalation and Indomethacin Challenge Study to Evaluate Safety, Tolerability and Pharmacokinetics of GSK4381406 in Healthy Participants
Brief Title: A First Time in Human Study to Evaluate the Safety and Tolerability of GSK4381406 in Healthy Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated prior to FSFV for strategic business reasons.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 218680
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Colitis, Ulcerative
Keywords: Gastrointestinal (GI); Intestinal permeability; First time in human (FTIH); Safety; Pharmacokinetics; Indomethacin challenge; Food effect
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Part 1: Cohort 1 - GSK4381406 or placebo (Experimental): Participants in Part 1 Cohort 1 will receive a single dose of GSK4381406 dose level 1 or placebo in Treatment Period 1 in fasted state, followed by GSK4381406 dose level 3 or placebo in Treatment Period 2 in fasted state with washout period of at least 40 days between each dose.
  Interventions: Drug: GSK4381406; Drug: Placebo
- Part 1: Cohort 2 - GSK4381406 or placebo (Experimental): Participants in Part 1 Cohort 2 will receive a single dose of GSK4381406 dose level 2 or placebo in Treatment Period 1 in fasted state, followed by GSK4381406 dose level 4 or placebo in Treatment Period 2 in fasted state with washout period of at least 40 days between each dose.
  Interventions: Drug: GSK4381406; Drug: Placebo
- Part 1: Cohort 3 - GSK4381406 or placebo (Experimental): Participants in Part 1 Cohort 3 will receive a single dose of GSK4381406 dose level 5 or placebo in Treatment Period 1 in fasted state, followed by GSK4381406 dose level 7 or placebo in Treatment Period 2 in fasted state with washout period of at least 40 days between each dose. Note: Requirement for Treatment Period 2 (dose level 7) will be determined by PK data of previous doses.
  Interventions: Drug: GSK4381406; Drug: Placebo
- Part 1: Cohort 4 - GSK4381406 or placebo (Experimental): Participants in Part 1 Cohort 4 will receive a single dose of GSK4381406 dose level 6 or placebo in Treatment Period 1 in fasted state, followed by GSK4381406 dose level 6 in Treatment Period 2 in fed state with washout period of at least 40 days between each dose.
  Interventions: Drug: GSK4381406; Drug: Placebo
- Part 2: Cohort 5 - GSK4381406 or placebo (Experimental): Participants in Part 2 Cohort 5 will receive 14 days of once daily repeat dosing of GSK4381406 dose level A or placebo in fasted state.
  Interventions: Drug: GSK4381406; Drug: Placebo
- Part 2: Cohort 6 - GSK4381406 or placebo (Experimental): Participants in Part 2 Cohort 6 will receive 14 days of once daily repeat dosing of GSK4381406 dose level B or placebo in fasted state.
  Interventions: Drug: GSK4381406; Drug: Placebo
- Part 2: Cohort 7 - GSK4381406 or placebo (Experimental): Participants in Part 2 Cohort 7 will receive 14 days of once daily repeat dosing of GSK4381406 dose level C or placebo in fasted state.
  Interventions: Drug: GSK4381406; Drug: Placebo
- Part 3 - GSK4381406 or Placebo and Indomethacin (Experimental): Participants in Part 3 will receive 3 days of once daily repeat dosing of GSK4381406 in Treatment Period 1 followed by placebo in Treatment Period 2, or placebo in Treatment Period 1 and GSK4381406 in Treatment Period 2 in a cross-over design with a washout period of at least 14 days between each dosing period. Participants will be dosed in fasted state. The participants will be challenged with indomethacin during the final 2 days of each dosing period.
  Interventions: Drug: GSK4381406; Drug: Placebo; Drug: Indomethacin

INTERVENTIONS:
Drug: GSK4381406 — GSK4381406 will be administered.
Drug: Placebo — Placebo will be administered.
Drug: Indomethacin — Indomethacin will be administered.
  Arms: Part 3 - GSK4381406 or Placebo and Indomethacin

SUMMARY:
This is a 3-part First Time in Human (FTIH) study to evaluate the safety, tolerability, and pharmacokinetics (PK) profile of GSK4381406 following administration of single ascending doses (Part 1), repeat ascending doses (Part 2), and repeat doses with an indomethacin challenge (Part 3) in healthy adult participants. Part 1 consists of 4 planned cohorts with up to 2 treatment periods in each and is expected to have 6 doses (but can accommodate up to 7 doses). The impact of food on PK of GSK4381406 will also be assessed. Part 2 will investigate 14 days of repeat dosing in 3 cohorts with 3 dose levels. Part 3 will evaluate the impact of repeat doses of GSK4381406 versus placebo on indomethacin induced changes in small intestinal permeability in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Body weight greater than (>)50 kg and body mass index (BMI) within the range 18-29.9 kilogram per meter square (kg/m^2) (inclusive)
* Male and female participants
* A female participant is eligible to participate if she is of non-childbearing potential
* Capable of giving signed informed consent

Exclusion Criteria:

* Medical history of cardiovascular, cerebrovascular (including transient ischemic attack (TIA), ischemic and hemorrhagic stroke), respiratory, hepatic, renal (including chronic kidney disease), gastrointestinal (including IBD and IBS), endocrine, hematologic (including anemia and coagulopathies), or neurological disorders
* Abnormal blood pressure (BP) (defined as systolic BP greater than or equal to [≥]130 millimetres of mercury (mmHg) or diastolic BP ≥85 mmHg) measured (based on the average of triplicate BP readings)
* Medical history of antihypertensive drugs
* Presence, or history within the past 14 days, of irregularities in bowel movements, including diarrhea (the passage of 3 or more loose or liquid stools per day) and constipation (3 or fewer bowel movements per week or requiring the use of laxatives).
* Symptomatic herpes zoster within 3 months prior to screening.
* Clinically significant multiple or severe drug allergies, intolerance to corticosteroids, or severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear immunoglobulin A [IgA] dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis).
* Any history or presence of malignancy except for basal cell or squamous epithelial carcinomas of the skin.
* Alanine transaminase (ALT) >1.5x Upper limit of normal (ULN)
* Total bilirubin >1.5x ULN (isolated total bilirubin >1.5xULN is acceptable if total bilirubin is fractionated and direct bilirubin lesser than [<]35 percentage [%]).
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (except for Gilbert's syndrome or asymptomatic gallstones).
* QT interval corrected for heart rate according to Fridericia's formula (QTcF) >450 millisecond (msec)
* Unable to refrain from the use of over-the-counter or prescription medication, including herbal medications and vitamins within 7 days or 5 half-lives (whichever is longer) prior to dosing until after follow-up visit, unless in the opinion of the Investigator and the GSK medical monitor, the medication will not interfere with the study procedures or compromise participant safety
* Use of a systemic antimicrobial within 30 days of screening
* The use of NSAIDs, including aspirin, are not permitted throughout the study (except on Part 3 Indomethacin challenge) and should not have been taken within 14 days immediately preceding the first dose of study intervention. For analgesia, paracetamol (acetaminophen) at doses of less than or equal to (≤)4 gram per day (g/day) is permitted
* Unable to refrain from consumption of red wine, Seville oranges, grapefruit, or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to first dose of study intervention until completion of the follow up period
* Live vaccine(s) within 1 month prior to screening or plans to receive such vaccines during the study
* Participation in the study would result in loss of blood or blood products in excess of 450 millilitre (mL) within the last 3 months prior to the Screening Visit. Blood donation during the study is not permitted
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day
* Current enrolment or past participation in another investigational study in which an investigational intervention (e.g., drug, vaccine, invasive device) was administered within the last 40 days or 5 half-lives, whichever is longer, before the first day of dosing (Day 1)
* Presence of Hepatitis B surface antigen (HBsAg) at screening or within 3 months prior to first dose of study intervention
* Positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention
* Positive hepatitis C ribo nucleic acid (RNA) test result at screening or within 3 months prior to first dose of study intervention.
* Positive pre-study drug/alcohol screen
* Regular use of known drugs of abuse, including tetrahydrocannabinol.
* Positive human immunodeficiency virus (HIV) antibody test.
* Evidence of active or latent tuberculosis (TB) as documented by medical history and examination, and TB testing: a positive (not indeterminate) TB test such as QuantiFERON-TB Gold Plus test
* Positive smoke breathalyzer levels indicative of smoking history at screening and each in-house admission to the clinical research unit or regular use of tobacco- or nicotine-containing products (e.g., nicotine patches or vaporizing devices) within 6 months prior to screening.
* Estimated glomerular filtration rate (eGFR) of <90 millilitre per minute per 1.73 meter square (mL/min/1.73 m^2) and / or UACR of >30 milligram per gram (mg/g) (>3 milligram per millimoles [mg/mmol]) at screening.
* Electrocardiogram (ECG) evidence of ischemic heart disease as determined by the Investigator.
* Positive test for Coronavirus disease 2019 (COVID-19) infection or signs and symptoms suggestive of COVID-19
* Regular excess alcohol consumption within 6 months prior to the study defined as an average weekly intake of >14 units for males and females
* Hypersensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study Additional exclusions for part 3 cohort only -
* Medical history of NSAIDs hypersensitivities, bronchial asthma, psychiatric and neurologic disorders, gastrointestinal disorders (including gastroesophageal reflux disease [GORD], gastritis, peptic ulcer disease and previous GI bleeding), cardiac or renal disease, coagulation defects and who are not on concomitant medication that may potentiate the potential harmful effects of indomethacin.
* Medical history of diabetes, defined as an HbA1c >5.6%, >39 mmol/mol.
* History of severe lactose intolerance or galactosaemia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-31 (Estimated); Primary Completion 2024-12-05 (Estimated); Study Completion 2024-12-05 (Estimated)

PRIMARY OUTCOMES:
Part 1 - Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to Day 40
Part 2 - Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to Day 54
Part 3 - Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to Day 34
Part 1 - Number of participants with clinically significant changes in hematology laboratory values | Up to Day 40
Part 2 - Number of participants with clinically significant changes in hematology laboratory values | Up to Day 54
Part 3 - Number of participants with clinically significant changes in hematology laboratory values | Up to Day 34
Part 1 - Number of participants with clinically significant changes in chemistry laboratory values | Up to Day 40
Part 2 - Number of participants with clinically significant changes in chemistry laboratory values | Up to Day 54
Part 3 - Number of participants with clinically significant changes in chemistry laboratory values | Up to Day 34
Part 1 - Number of participants with clinically significant changes in urinalysis | Up to Day 40
Part 2 - Number of participants with clinically significant changes in urinalysis | Up to Day 54
Part 3 - Number of participants with clinically significant changes in urinalysis | Up to Day 34
Part 1 - Number of participants with clinically significant changes in vital signs | Up to Day 40
Part 2 - Number of participants with clinically significant changes in vital signs | Up to Day 54
Part 3 - Number of participants with clinically significant changes in vital signs | Up to Day 34
Part 1 - Number of participants with clinically significant changes in 12-lead Electrocardiogram (ECG) readings | Up to Day 40
Part 2 - Number of participants with clinically significant changes in 12-lead Electrocardiogram (ECG) readings | Up to Day 54
Part 3 - Number of participants with clinically significant changes in 12-lead Electrocardiogram (ECG) readings | Up to Day 34

SECONDARY OUTCOMES:
Part 1 - Area under the plasma concentration-time curve (AUC) from time zero to 24-hour post-dose [AUC(0-24) | Up to 24 hours post dose
Part 1 - AUC from time zero to last quantifiable concentration [AUC(0-t) | Up to Day 40
Part 1 - AUC from time zero to infinity [AUC(0-inf) | Up to Day 40
Part 1 - Maximum observed plasma drug concentration (Cmax) | Up to Day 40
Part 1 - Time to maximum observed plasma drug concentration (tmax) | Up to Day 40
Part 1 - Time of last quantifiable concentration (tlast) | Up to Day 40
Part 1 - Apparent terminal phase half-life (t½) | Up to Day 40
Part 2 - AUC from time zero to last quantifiable concentration [AUC(0-t) | Day 1 and Day 14
Part 2 - AUC over the dosing interval [AUC(0-tau) | Day 1 and Day 14
Part 2 - Maximum observed plasma drug concentration (Cmax) | Day 1 and Day 14
Part 2 - Time to maximum observed plasma drug concentration (tmax) | Day 1 and Day 14
Part 2 - AUC from time zero to infinity [AUC(0-inf) | Day 14 to Day 54
Part 2 - Apparent terminal phase half-life (t½) | Day 14 to Day 54
Part 2 - Pre-dose (trough) plasma concentrations (Ctau) | Day 1 to Day 14
Part 2 - Accumulation ratios for Cmax (R) | Day 1 and Day 14
Part 2 - Accumulation ratios for AUC(0-tau) (Ro) | Day 1 and Day 14
Part 1: Cohort 4 - AUC from time zero to infinity [AUC(0-inf) | Up to Day 40
Part 1: Cohort 4 - Maximum observed plasma drug concentration (Cmax) | Up to Day 40
Part 1: Cohort 4 - Time to maximum observed plasma drug concentration (tmax) | Up to Day 40
Part 3 - Lactulose:rhamnose ratio over 0-5 hour in urine | At Day 1, 3, 17 and 20
  Lactulose and rhamnose concentrations in urine will be collected over 0-2 hour and 2-5 hour, which will be used to derive the ratio over 0-5 hour

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/